CLINICAL TRIAL: NCT03936712
Title: Effects of Energy Drink on Performance and Psycho-Physiological Response to Physical Exercise
Brief Title: Effect of Energy Drink on Sport Performance and Psycho-Physiological Responses.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Higher Institute of Sport and Physical Education of Sfax (Other)
Responsible Party: Principal Investigator, Ammar Achraf, Principal Investigator, The Higher Institute of Sport and Physical Education of Sfax
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Hamdi Chtourou
Record Dates: First submitted 2019-04-24; First posted 2019-05-03 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Physical Activity
Keywords: Energy drinks; Exercise; Physiological response; Mood State; Fatigue
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Energy Drinks

STUDY DESIGN:
Intervention Model Description: A double blind, placebo-controlled, and counterbalanced crossover design was used for this work
Who Masked: Participant
Masking Description: To avoid identification, two opaque and unmarked cans [24-26] of Red Bull or Placebo were ingested by each participant (i.e., 500 mL) in the presence of a researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red Bull drink (RB) (Experimental): Over the study, three participants were unable to complete all test sessions due to muscle pain or injury . Thus, 19 participants (age: 21.2±1.2 years; height: 1.76±0.8 m; body-mass: 76.6±12.6 kg) completed all test sessions
  Interventions: Dietary Supplement: Energy Drink
- Placebo drink (Placebo Comparator): 19 participants (age: 21.2±1.2 years; height: 1.76±0.8 m; body-mass: 76.6±12.6 kg)
  Interventions: Dietary Supplement: Placebo Drink

INTERVENTIONS:
Dietary Supplement: Energy Drink — Each participant visited the laboratory for two formal test sessions, drinking a caffeine-containing ED (RB) and a caffeine and taurine free beverage drink (PL). All sessions were arranged in the early evening hours to avoid any time of day effects. The two definitive test sessions were separated by an interval of seven days to allow sufficient recovery between tests and to ensure caffeine washout. To avoid identification, two opaque and unmarked cans of RB or PL were ingested by each participant (i.e., 500 mL) in the presence of a researcher. The two drinks were similar in volume, texture, and appearance. One can of RB drink (i.e., 250ml) contained 80 mg of caffeine, 1 g of taurine, 27 g of carbohydrates, 0.6 g of protein, 5 mg vitamin B6 and 487 kJ of energy.
  Arms: Red Bull drink (RB)
Dietary Supplement: Placebo Drink — The PL drink was prepared by an agri-food engineer; it did not contain any caffeine or taurine, but comprised carbonated water, carbohydrates, citric acid lemon juice reconstituted from concentrate (1 %), supplemented by flavorings, of sodium citrate, acesulfame K, sucralose, potassium sorbate and RB (a flavoring that contains propylene glycol E1520 (0.23 mL).
  Arms: Placebo drink

SUMMARY:
This work aimed to examine the effects of drinking an "energy drink" upon (i) short-term maximal performance, (ii) reaction times and (iii) psychological factors (i.e., mood state, ratings of perceived exertion (RPE) and affective load) and on physiological parameters such as blood pressure, blood glucose, hematological parameters and other biochemical parameters.

DETAILED DESCRIPTION:
A total of 22 healthy and regularly active physical-education male students from various sports disciplines volunteered to participate in this study. Potential participants were initially screened through telephone interviews based on the inclusion criteria: 18-40 years of age, BMI less than 25 kg/m2, and low (<1.5g/month ) and not regular caffeine users. Exclusion criteria included diagnosis of any chronic metabolic disease such as type 2 diabetes or cardiovascular disease, an auto-immune disease such as rheumatoid arthritis, lupus or type 1 diabetes, liver disease and the intake of any medications/ or dietary supplements known to influence blood glucose concentrations and/or blood pressures.

The study was conducted according to the declaration of Helsinki and the protocol was fully approved (identification code: 8/16) by the review board "Local committee of the Laboratory of Biochemistry, CHU Habib Bourguiba, Sfax, Tunisia." After a throughout explanation of the protocol and responses to all questions, participants signed a written informed consent.

Subjects were instructed to avoid nicotine, alcohol, dietary supplements, medications and all other stimulants and to maintain their normal dietary, sleep and physical activity patterns before test sessions. Caffeine and other caffeinated products (e.g., chocolate, caffeinated gums, caffeine containing beverages) were avoided for 48 hours and food for at least 4 hours before testing.

A double blind, placebo-controlled, counterbalanced, crossover design was adopted for this study. The randomized order of testing was determined using free online software (www.randomization.com). Neither staff nor participants were informed about the names of the two drinks, and blinding was strictly maintained by emphasizing to both staff and participants that both drinks adhered to healthy principles, and that each was advocated by certain sports medicine experts. Two familiarization sessions were completed before definitive test sessions in order to eliminate any learning effects on physical performance and reaction time measurements. During the second familiarization session, body mass and height were recorded. Each participant visited the laboratory for two formal test sessions, drinking a caffeine-containing ED (RB) and a caffeine and taurine free beverage drink (PL). All sessions were arranged in the early evening hours to avoid any time of day effects. The two definitive test sessions were separated by an interval of seven days to allow sufficient recovery between tests and to ensure caffeine washout. To avoid identification, two opaque and unmarked cans of RB or PL were ingested by each participant (i.e., 500 mL) in the presence of a researcher. The two drinks were similar in volume, texture, and appearance. One can of RB drink (i.e., 250ml) contained 80 mg of caffeine, 1 g of taurine, 27 g of carbohydrates, 0.6 g of protein, 5 mg vitamin B6 and 487 kJ of energy. The PL drink was prepared by an agri-food engineer; it did not contain any caffeine or taurine, but comprised carbonated water, carbohydrates, citric acid lemon juice reconstituted from concentrate (1 %), supplemented by flavorings, of sodium citrate, acesulfame K, sucralose, potassium sorbate and RB (a flavoring that contains propylene glycol E1520 (0.23 mL).

Beverages were prepared, shaken and chilled in a refrigerator at 14h00 by an investigator who took no part in the test sessions or data analysis, but prepared the alphanumeric code identifying the tested drink. At 17h00, the cooled beverages were served in sealed plastic opaque water bottles and consumed using an opaque straw. Participants were instructed to drink the fluid quickly (within 1±0.5 min) 60 minutes before their test session and not to discuss or compare tastes or to make any assumptions about what they had ingested. The interval of 60 minutes was chosen as optimal for a complete caffeine absorption and thus a peaking of a caffeine concentration .

Subjects were supervised by staff to ensure that they drank the entire quantity of fluid, and no exchange of bottles was allowed. The last standardized meal (i.e., lunch) before the beginning of the test session was taken at 13h00. Temperature and relative humidity of the laboratory were similar over the test sessions, with a temperature of around 22°C and a relative humidity between 45 and 55 %. During each test session (from 18h00), resting blood glucose and blood pressures were measured and the participants completed the POMS questionnaire.

A 5-min treadmill warm-up was performed. After that, the reaction time, and handgrip force were determined, and the 30-s Wingate test was performed. RPE scores, blood glucose and blood pressures were then measured, and the affective load was calculated. To investigate the effects of RB on the acute physiological and psychological responses to exercise, blood measures and psychological test measures were collected immediately pre- and post-exercise.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age,
* BMI less than 25 kg/m2,
* low (<1.5g/month [20]) caffeine users
* not regular caffeine users.

Exclusion Criteria:

* chronic metabolic disease such as type 2 diabetes and cardiovascular disease
* auto-immune disease such as rheumatoid arthritis, lupus or type 1 diabetes,
* liver disease
* intake of any medications/ or dietary supplements known to influence blood glucose and/or blood pressures.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-01-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Change in Wingate-test physical performance from PL to RB condition | The performance in Wingate test was measured 1 hour following the consumption of supplementations in the first and second test sessions (RB session and PLA session) to assess possible beneficial effect of RB supplementation in physical performance
  A calibrated mechanically-braked cycle ergometer (Monark 894; Stockholm, Sweden) interfaced with a microcomputer was utilized for the 30-s Wingate test. Subjects pedaled as fast as possible for 30-s against a constant load calculated according to the participant's body-mass (i.e., 8.7%). After maintaining a constant ~60rpm speed for 4-6-s against minimal resistance, the selected load was applied. The participant sat on the cycle throughout and was strongly encouraged to maximize pedaling rates and to maintain a high speed. Peak and mean power (i.e., average of power output the 30-s) were recorded. The fatigue index was calculated as follows:
  Fatigue index (%) = [(peak power-minimal power)/ peak power×100]. The ICC and SEM showed excellent reliability for peak power (ICC>0.98, absolute SEM <0.21), mean power (ICC>0.98, absolute SEM <0.23) and fatigue index (ICC>0.76, absolute SEM <1.99).
Change in Reaction Time Performance from PL to RB condition | The reaction time performance was measured 1 hour following the consumption of supplementations in the first and second test sessions (RB session and PLA session) to assess possible beneficial effect of RB in reaction time performance
  A simple visual reaction time test assessed alertness and motor reaction-speed. Subjects responded as quickly as possible to presentation of a stimulus (the image of a black box) on a computer screen (15" LCD). When this appears, the participant should press the index finger on a computer key. The signal appeared in random order within 1-10-s time intervals. Each participant was allowed ten attempts and the mean reaction time was calculated, using React! V0.9 software.The ICC and SEM showed excellent reliability for reaction time (ICC>0.89, absolute SEM <0.14) measurement.
Change in Strength Physical Performance (i.e., Handgrip) from PL to RB condition | Handgrip performance was measured 1 hour following the consumption of supplementations in the first and second test sessions (RB session and PLA session) to assess possible beneficial effect of RB supplementation in strength (i.e., Handgrip) performance
  Handgrip strength was recorded by dynamometer (T.K.K. 5401; Takei, Tokyo, Japan). The maximal handgrip force was determined for the dominant hand. Participants exerted their maximal strength for 4-5-s. With the hand hanging downwards, the dynamometer was
Change in Rating of Perceived Exertion (RPE) and Affective Load from PL to RB condition | RPE and Affective Load were measured immediately following the first and second training sessions (RB and PL sessions) to assess any beneficial effect of the consumed RB (1 hour before session) on fatigue and load perception
  The original Borg RPE scale rates exertion subjectively during or after physical exercise on a 15-point scale ranging from six (very very light) to twenty (very very hard). It was used to calculate the affective load; the affective load was obtained as the difference between the perceived exertion (negative affective response) and pleasure scores (positive affective response). For example, with an RPE score of six, the negative affective response is zero and the positive affective response is -14. However, if the RPE score rises to 20, the negative affective response is +14 and the positive affective response is zero. The potential affective load thus ranges from -14 to +14. A negative affective load score indicates the dominance of pleasant affective responses and a positive affective load represents the dominance of unpleasant affective responses.
Change in Mood States (POMS) from PL to RB condition | POMS was measured immediately following the first and second training sessions (RB and PL sessions) to assess any beneficial effect of the consumed RB (1hour before session) on perception of tension, depression, anger, vigor, fatigue, and confusion
  The evaluation of mood states used the French language version of the POMS questionnaire. Responses to 65 adjectives (ranging from "Zero" (i.e., not at all) to "Four" (i.e., extremely) assessed immediate mood states in seven dimensions: tension, depression, anger, vigor, fatigue, confusion and interpersonal relationships.
Change in Blood pressure and blood glucose from pre- to post-training session using RB condition | Blood pressure and blood glucose were measured 1 hour after RB supplementation (correspond to pre-training session) and also immediately following the training session to assess any exercise effect on blood pressure/glucose responses during RB condition
  Blood glucose was measured using the electrochemical sensor Rightest GM260 Blood Glucose Monitoring System (Bionime Corporation, Taichung City, Taiwan). The finger tip was pricked with a lancing device, and a specific test strip was soaked with blood was inserted into the measuring apparatus, with an estimate appearing within 5 seconds. Blood pressure was measured by the same physician using a stethoscope (Spengler, Germany) and sphygmomanometer (Spengler, Germany).
Change in Blood pressure and blood glucose from pre- to post-training session using PL condition | Blood pressure and blood glucose were measured 1 hour after PL supplementation (correspond to pre-training session) and also immediately following the training session to assess any exercise effect on blood pressure/glucose responses during PL condition
  Blood glucose was measured using the electrochemical sensor Rightest GM260 Blood Glucose Monitoring System (Bionime Corporation, Taichung City, Taiwan). The finger tip was pricked with a lancing device, and a specific test strip was soaked with blood was inserted into the measuring apparatus, with an estimate appearing within 5 seconds. Blood pressure was measured by the same physician using a stethoscope (Spengler, Germany) and sphygmomanometer (Spengler, Germany).
Change in hematological parameters from pre- to post-training session using RB condition | Hematological parameters were measured 1 hour after RB supplementation (correspond to pre-training session) and also immediately following the training session to assess any exercise effect on hematological responses during RB condition
  Haematological parameters (i.e., white blood cells (WBC), neutrophils (NEU), red blood cells (RBC), hemoglobin (HGB), hematocrit (HCT)and platelets (PLT) were determined using a multichannel automated blood cell analyser Beckman Coulter Gen system-2 (Coulter T540)
Change in hematological parameters from pre to post training session using PL condition | Hematological parameters were measured 1 hour after PL supplementation (correspond to pre-training session) and also immediately following the training session to assess any exercise effect on hematological responses during PL condition
  Haematological parameters (i.e., white blood cells (WBC), neutrophils (NEU), red blood cells (RBC), hemoglobin (HGB), hematocrit (HCT)and platelets (PLT) were determined using a multichannel automated blood cell analyser Beckman Coulter Gen system-2 (Coulter T540)
Change in muscle damage parameters from pre to post training session using RB condition | Muscle damage parameters were measured 1 hour after RB supplementation (correspond to pre-training session) and also immediately following the training session to assess any exercise effect on muscle damage responses during RB condition
  muscle damage markers: Creatinine kinase (CK), Alkaline phosphate (PAL), Gammaglutamyl (GGT), Lactate dehydrogenase (LDH), and c-reactive protein (CRP) were determined spectrophotometrically using Abott Architect Ci 4100.
Change in muscle damage parameters from pre to post training session using PL condition | Muscle damage parameters were measured 1 hour after PL supplementation (correspond to pre-training session) and also immediately following the training session to assess any exercise effect on muscle damage responses during PL condition
  muscle damage markers: Creatinine kinase (CK), Alkaline phosphate (PAL), Gammaglutamyl (GGT), Lactate dehydrogenase (LDH), and c-reactive protein (CRP) were determined spectrophotometrically using Abott Architect Ci 4100.
Change in oxidative stress parameters from pre to post training session using RB condition | Oxidative stress parameters were measured 1 hour after RB supplementation (correspond to pre-training session) and also immediately following the training session to assess any exercise effect on oxidative stress responses during RB condition
  Oxididative stress response (i.e., malondialdehyde (MDA), superoxide dismutase (SOD), glutathione peroxidase (GPx), Catalase (CAT), uric acid (UA)) and c-reactive protein (CRP)) were determined spectrophotometrically using Abott Architect Ci 4100.
Change in oxidative stress parameters from pre to post training session using PL condition | Oxidative stress parameters were measured 1 hour after PL supplementation (correspond to pre-training session) and also immediately following the training session to assess any exercise effect on oxidative stress responses during PL condition
  Oxididative stress response (i.e., malondialdehyde (MDA), superoxide dismutase (SOD), glutathione peroxidase (GPx), Catalase (CAT), uric acid (UA)) and c-reactive protein (CRP)) were determined spectrophotometrically using Abott Architect Ci 4100.

IPD SHARING:
Plan to Share IPD: No